CLINICAL TRIAL: NCT02725255
Title: Design and Clinical Evaluation of a School Meal With Deworming Properties
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kenya Medical Research Institute (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Elijah M. Songok, Prof. Elijah M. Songok, Kenya Medical Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSC2580
Record Dates: First submitted 2016-02-28; First posted 2016-03-31 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Helminthiasis; Tinea Capitis; Anemia
MeSH Terms: conditions — Helminthiasis; Tinea Capitis; Anemia | interventions — Albendazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Papaya seed porridge (Experimental): Arm receiving porridge fortified with dried papaya seeds (Ujiplus)
  Interventions: Dietary Supplement: Ujiplus
- Albendazole and Plain porridge (Active Comparator): Arm receiving the approved albendazole treatment of 400mg once with plain porridge daily (without papaya seeds)
  Interventions: Drug: Albendazole
- Plain porridge (Placebo Comparator): arm receiving 300ml plain porridge daily (without papaya seeds)
  Interventions: Dietary Supplement: uji

INTERVENTIONS:
Dietary Supplement: Ujiplus — Maize flour fortified with micronutrients and dried ground papaya (Carica papaya) seeds. The flour was used to prepare porridge and each child given a serving of 300 ml every school day for 60 days.
  Arms: Papaya seed porridge
Drug: Albendazole — 400mg of albendazole given to each child once at the beginning of the study and maize flour porridge fortified only with micronutrients cooked and served to each child, 300ml per day for 60 days.
  Other Names: Albenza
  Arms: Albendazole and Plain porridge
Dietary Supplement: uji — maize flour porridge fortified only with micronutrients, cooked and served to each child 300ml per day for 60 days.
  Arms: Plain porridge

SUMMARY:
Intestinal parasites (IP) are among the world's neglected tropical diseases. Morbidity due to IPs is greatest in school-age children who typically have the highest burden of infection. In 2001, WHO passed a resolution for the use of large-scale mass drug administration (MDA) of antihelminthic drugs to deworm children in developing countries. Though initially effective, there is concern that MDA might not be sustainable over extended periods especially considering the large children populations and the high frequency of dosing. Further, the MDAs exert increasing drug pressure on parasite populations, a circumstance that is likely to favor parasite genotypes that can resist anthelmintic drugs. There is hence a need for alternatives that are not only affordable and sustainable but easier to implement in the long term with a minimal chance of development of resistance. The investigators propose to develop and test the feasibility of a corn porridge meal fortified with papaya fruit extracts that have been shown to have antihelminthic properties. The investigators intend to evaluate its efficacy when given through school feeding programs and compare the outcome with albendazole- the recommended MDA agent for deworming school children. The investigators will design and formulate the product and test it among children in three primary schools in Western Kenya.

DETAILED DESCRIPTION:
Background: Soil transmitted helminthes (STHs) are among the world's neglected tropical diseases. Morbidity due to STHs is greatest in school-age children who typically have the highest burden of infection. In 2001, WHO passed a resolution for the use of large-scale mass drug administration (MDA) to deworm vulnerable children. Though effective, there is concern that MDA might not be sustainable over extended periods. Additionally the current MDA strategy do not consider child malnutrition, a very common malady in resource limited countries. The investigators report a pilot evaluation of an innovation that bundles school feeding and deworming.

The investigators designed a maize (corn) flour fortified with grounded dried papaya (Carica papaya) seeds and used it to prepare porridge as per the usual school meal recipe. Children from three primary schools from Nandi County in Kenya were randomized into three arms: One school received 300 ml papaya fortified porridge daily (test school), a second school received similar serving of plain porridge without the pawpaw ingredient (placebo) and a third school received the placebo porridge and the conventional MDA approach of one time 400mg dosage of albendazole. Prior to the randomization, an initial baseline stool microscopy analysis was done to determine presence and intensity of intestinal worms. Core indicators of nutrition-height, weight and hemoglobin counts-were also assessed. The children were monitored daily for two months and final stool sample analysis and clinical monitoring done at the end of the study. Baseline and follow-up data were analyzed and compared through SAS version 9.1 statistical package.

ELIGIBILITY:
Inclusion Criteria:

* Consenting parents and guardians

Exclusion Criteria:

* children with known allergy to papaya fruit products

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 326 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
parasite egg count | 60 days after randomization
  ova and cyst counts of various helminths in stool sample at end of intervention

SECONDARY OUTCOMES:
Body Mass Index for age | 60 days after intervention
  Height, Weight and age were collected. BMI was calculated using WHO guidelines.
school attendance | 60 days after randomization
  school register used to gather information of attendance, enrollment and retention of students
haemoglobin levels | baseline and after 60 days
  blood sample is taken for hemoglobin amounts at start and end of intervention
Number of children with tinea capitis | 60 days after randomization
  Number of children with tinea capitis (ringworms) 60 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Elijah M Songok, PhD, Principal Investigator — Kenya Medical Research Institute

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Okeniyi JA, Ogunlesi TA, Oyelami OA, Adeyemi LA. Effectiveness of dried Carica papaya seeds against human intestinal parasitosis: a pilot study. J Med Food. 2007 Mar;10(1):194-6. doi: 10.1089/jmf.2005.065. PMID 17472487
- [Background] Kermanshai R, McCarry BE, Rosenfeld J, Summers PS, Weretilnyk EA, Sorger GJ. Benzyl isothiocyanate is the chief or sole anthelmintic in papaya seed extracts. Phytochemistry. 2001 Jun;57(3):427-35. doi: 10.1016/s0031-9422(01)00077-2. PMID 11393524
- [Background] Ash LR, Orihel TC, Savioli L. Bench aids for the diagnosis of intestinal parasites. Geneva. World Health Organization, 1994
- [Background] Sapaat A, Satrija F, Mahsol HH, Ahmad AH. Anthelmintic activity of papaya seeds on Hymenolepis diminuta infections in rats. Trop Biomed. 2012 Dec;29(4):508-12. PMID 23202594
- [Derived] Kugo M, Keter L, Maiyo A, Kinyua J, Ndemwa P, Maina G, Otieno P, Songok EM. Fortification of Carica papaya fruit seeds to school meal snacks may aid Africa mass deworming programs: a preliminary survey. BMC Complement Altern Med. 2018 Dec 7;18(1):327. doi: 10.1186/s12906-018-2379-2. PMID 30526582